CLINICAL TRIAL: NCT04047901
Title: Effect of Physical Training in Patients With Heart Failure Caused by Chemotherapy for Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other); Cancer Institute of Sao Paulo (Unknown); Hospital Sirio-Libanes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC COP 002/15/002
Record Dates: First submitted 2019-03-29; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-03

CONDITIONS: Insufficiency;Cardiac; Cancer; Cardiotoxicity; Heart Failure
Keywords: autonomic dysfunction; baroreflex control; ergorreflex control; muscle myopaty
MeSH Terms: conditions — Heart Failure; Neoplasms; Cardiotoxicity; Primary Dysautonomias | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): A group of patients who will not be trained will be evaluated at baseline (pre) and after 16 weeks.
  They are oriented to maintain lifestyle changes
- Training group (Experimental): Patients will complete 16 weeks of training including 40 minutes of aerobic training, 15 minutes of resistive exercise and 5 minutes of relaxation.
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — Patients undergo 16 weeks of physical training
  Arms: Training group

SUMMARY:
New therapies for cancer increased patient survival, but led to the recognition of adverse effects associated with cancer treatment, such as the use of chemotherapy. Cardiotoxicity is the most significant adverse effect, which affect the functional capacity and quality of life and is associated with high morbidity and mortality, regardless of the oncological prognosis. One of the manifestations of cardiotoxicity is ventricular dysfunction that can lead to heart failure. Neuro humoral hyperactivation with increased sympathetic nerve activity is a typical manifestation of heart failure and is associated with worse prognosis. Studies have shown that physical training significantly reduces sympathetic nerve activity in addition to improving muscle blood flow, reversing effects on skeletal muscle and improving quality of life. The hypothesis is that physical training may reduce sympathetic nerve activity and vasoconstrictor status in patients with heart failure caused by anthracyclines, as well as improving baroreflex and chemoreflex sensibility, mechanoreflex and metaborreflex control and skeletal myopathy.

DETAILED DESCRIPTION:
The investigators included patients> 18 years, left ventricular ejection fraction <= 0.55, functional class (NYHA) I-III, under medical treatment for heart failure. Patients with coronary artery disease, moderate to severe valve disease, positive Chagas serology, inability to participate in an exercise program are excluded.

Primary outcome: Muscle sympathetic nerve activity Secondary outcome: arterial baroreflex sensitivity, peripheral chemorreflex sensitivity, mecanic and muscuclar metaborreflex control, ubiquitin proteasome system activity.

Patients were divided into 2 groups-trained (n = 10) and non-trained (n = 10). Patients in the trained group will complete 16 weeks of aerobic training. Evaluation of cardiac function, functional capacity, quality of life and biochemical evaluation (troponin, hs-CRP and BNP). For muscle evaluation will be performed biopsy of the vastus lateralis muscle

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old
* Funcional Class I-III (NYHA)
* Ejection fraction < o,55
* treated for heart failure

Exclusion Criteria:

* Coronary artery disease
* Moderate to major valve disease
* Positive serology for Chagas
* Inability to perform physical exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11-07 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Measure muscular sympathetic nervous activity | 16 weeks
  The sympathetic nervous activity is assessed by the microneurography technique

SECONDARY OUTCOMES:
Evaluate baroreflex activity | 16 weeks
  Evaluation of muscular sympathetic nervous activity at rest by the technique of microneurography, evaluation of the muscular blood flow by venous occlusion plethysmography technique
Evaluate quimiorreflex sensibility | 16 weeks
  Evaluation of muscular sympathetic nervous activity at rest by the technique of microneurography, evaluation of the muscular blood flow by venous occlusion plethysmography technique
Evaluate Mecanorreflex control | 16 weeks
  Evaluation of muscular sympathetic nervous activity at rest by the technique of microneurography, evaluation of the muscular blood flow by venous occlusion plethysmography technique
Evaluate metaborreflex control | 16 weeks
  Evaluation of muscular sympathetic nervous activity at rest by the technique of microneurography, evaluation of the muscular blood flow by venous occlusion plethysmography technique
Evaluation of skeletal myopathy | 16 weeks
  muscle biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute of University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No